CLINICAL TRIAL: NCT00036361
Title: Broad Effectiveness: Study With Aripiprazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-087
Record Dates: First submitted 2002-05-08; First posted 2002-05-10 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is effective in the treatment of a large number of persons diagnosed with schizophrenia or schizoaffective disorders

ELIGIBILITY:
* Patients with Schizophrenia or Schizoaffective Disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444
Dates: Start 2002-07; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Safety Assessments

SECONDARY OUTCOMES:
Safety Assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Wallingford, Connecticut, United States